CLINICAL TRIAL: NCT00680342
Title: A Multicenter, Randomized, Double-masked, Placebo-controlled Phase II Study to Assess the Safety and Efficacy of a Standardized Orally Administered Silymarin Preparation (Legalon) for the Treatment of Patients With Chronic Hepatitis C Who Failed Conventional Antiviral Therapy
Brief Title: Phase II Trial of Silymarin for Patients With Chronic Hepatitis C Who Have Failed Conventional Antiviral Treatment
Acronym: SyNCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pennsylvania (Other); University of North Carolina, Chapel Hill (Other); Thomas Jefferson University (Other); Beth Israel Deaconess Medical Center (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01AT003566 (NIH); IND 74,887
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Silymarin; milk-thistle extract; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo (lactose pill)
  Interventions: Other: Placebo
- 2 (Experimental): 700mg of Legalon (silymarin) three times daily
  Interventions: Drug: Silymarin
- 3 (Experimental): 420mg Legalon (silymarin) three times daily
  Interventions: Drug: Silymarin

INTERVENTIONS:
Drug: Silymarin — 700mg dose (5 pills, three times daily) for 24-week treatment period
  Other Names: Legalon; milk thistle
  Arms: 2
Drug: Silymarin — 420mg dose (5 pills, three times daily) for 24-week treatment period
  Other Names: Legalon; milk thistle
  Arms: 3
Other: Placebo — Placebo (5 pills, three times daily) for 24-week treatment period
  Other Names: lactose pill
  Arms: 1

SUMMARY:
Silymarin (Legalon), also known as milk thistle, is an alternative medicine commonly found in health food and vitamin stores. People with liver disease sometimes use silymarin because it is thought to have liver protecting effects; however, this benefit has not been proven. The purpose of this research study is to determine the effectiveness of silymarin and assess the safety of different silymarin doses in patients with varying severity of liver disease compared to a placebo (lactose pill).

Eligible subjects will be randomized to treatment with placebo or one of two dosages of Legalon® 420 mg or 700 mg administered orally thrice daily. Investigators and subjects will be masked to treatment assignment. The study design includes a screening period during which patients will undergo full medical evaluation to verify protocol eligibility and a treatment period of 24 weeks during which time clinic visits and laboratory studies will be performed every 2-4 weeks to monitor for safety and efficacy of therapy. Subjects will continue to be followed for an additional 12 weeks after the completion of study medication to monitor for adverse events and investigate post-treatment outcomes. Participation in this research study requires the subject to travel to the clinic for at least 10 visits so recruitment will be limited to a geographically restricted area around participating clinical centers.

DETAILED DESCRIPTION:
This proposal is a phase II study that will evaluate the safety and efficacy of silymarin for the treatment of subjects with chronic hepatitis C who did not respond to conventional antiviral therapy. The primary objectives of this study are to assess the safety and adverse event profile of silymarin over a range of doses compared to placebo and to assess efficacy of silymarin in normalizing serum aminotransferase activity in patients with chronic hepatitis C. Secondary objectives are to characterize the effect of silymarin on serum levels of HCV RNA and to explore relationships between silymarin therapy and serum biomarkers of HCV hepatic disease activity (oxidative stress, apoptosis, and fibrogenesis).

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years at screening.
* Serum HCV RNA above quantifiable level of detection by any assay after the end of previous therapy.
* ALT > 65 IU/L (i.e., approximately 1.5 X upper limit of normal) obtained during the screening period.
* Previous treatment with any interferon-based therapy without sustained virological response.
* Negative urine pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of silymarin. Females of childbearing potential must be using two reliable forms of effective contraception during the study (while on drug and during follow-up).

Exclusion Criteria:

* Use of silymarin or other milk thistle preparations within 30 days prior to screening.
* Use of other antioxidants such as vitamin E, vitamin C, glutathione, alpha-tocopherol, or non-prescribed complementary alternative medications (including dietary supplements, megadose vitamins, herbal preparations, and special teas) within 30 days prior to screening. A multivitamin at standard doses will be allowed.
* Use of silymarin or other antioxidants or non-prescribed complementary alternative medications (as above) during the screening period or patient unwilling to refrain from taking these medications through completion of the study.
* Any antiviral therapy within 6 months prior to screening visit.
* Known allergy/sensitivity to milk thistle or its preparations.
* Evidence of poorly-controlled diabetes (defined as HbA1c > 8% in patients with diabetes).
* Use of warfarin, metronidazole or acetaminophen (greater than two grams per day) within 30 days of screening.
* Lactose intolerance defined as patient reported inability to tolerate milk products.
* Previous liver biopsy that demonstrated presence of moderate to severe steatosis or evidence of steatohepatitis.
* Positive test for anti-HIV or HBsAg within 5 years of screening.
* Average alcohol consumption of more than one drink or equivalent (>12 grams) per day or more than two (2) drinks on any one day over the 30 days prior to screening. Patients who met either criterion more than 30 days ago must have consumed a monthly average of 12 grams or less per day of alcohol for at least six months prior to screening.
* History of other chronic liver disease, including metabolic diseases, documented by appropriate test(s).
* Women with ongoing pregnancy or breast-feeding, or contemplating pregnancy.
* Serum creatinine level 2.0 mg/dL or greater at screening or CrCl ≤ 60cc/min, or currently on dialysis. The creatinine clearance (CrCl) will be calculated according to Cockcroft-Gault.
* Evidence of drug abuse within 6 months prior to screening or during the screening period.
* Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dl, total bilirubin > 1.5 mg/dl, or PT/INR > 1.3 times normal at screening, or history or presence of ascites or encephalopathy, or bleeding from esophageal varices.
* History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, or active gastrointestinal conditions that might interfere with drug absorption).
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hepatitis, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis) that could affect inflammatory biomarkers.
* History of solid organ or bone marrow transplantation.
* History of thyroid disease poorly controlled on prescribed medications.
* Use of oral steroids for more than 14 days within 30 days prior to screening.
* Participation in a research drug trial, exclusive of the SyNCH Phase I trial, within 6 months of enrollment.
* Inability or unwillingness to provide informed consent or abide by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Efficacy - whether or not serum ALT (mg/dl) is less than or equal to 45 IU/L (approximate normal range) or achieves at least 50% decline to less than 65 IU/L (approximately 1.5 times the upper limit of normal) | 24-week treatment period
Safety - occurence of a dose-limiting toxicity | 24-week treatment period

SECONDARY OUTCOMES:
Adherence - summary of missed dose information obtained from patient diaries and dose counts | 24 week treatment period
Biomarkers - the following relationships will be explored: dose and change in biomarkers, changes in biomarkers and rate of treatment success, change in biomarkers and rate of toxicity | 24 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fried, MD, Principal Investigator — University of North Carolina, Chapel Hill; Victor Navarro, MD, Principal Investigator — Thomas Jefferson University; Nezam Afdhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center; K. Rajender Reddy, MD, Principal Investigator — University of Pennsylvania; Steven Belle, PhD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Reddy KR, Belle SH, Fried MW, Afdhal N, Navarro VJ, Hawke RL, Wahed AS, Doo E, Meyers CM; SyNCH Study Group. Rationale, challenges, and participants in a Phase II trial of a botanical product for chronic hepatitis C. Clin Trials. 2012 Feb;9(1):102-12. doi: 10.1177/1740774511427064. Epub 2011 Nov 4. PMID 22058086
- [Result] Fried MW, Navarro VJ, Afdhal N, Belle SH, Wahed AS, Hawke RL, Doo E, Meyers CM, Reddy KR; Silymarin in NASH and C Hepatitis (SyNCH) Study Group. Effect of silymarin (milk thistle) on liver disease in patients with chronic hepatitis C unsuccessfully treated with interferon therapy: a randomized controlled trial. JAMA. 2012 Jul 18;308(3):274-82. doi: 10.1001/jama.2012.8265. PMID 22797645